CLINICAL TRIAL: NCT04909229
Title: Randomized Controlled Trial Examining Real-World Effectiveness of a Prescription Digital Therapeutic for the Treatment of Insomnia
Brief Title: Prescription Digital Therapeutic for the Treatment of Insomnia
Acronym: SLEEP-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Mayo Clinic (Other); National Evaluation System for health Technology Coordinating Center (Other); Pear Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000029050
Record Dates: First submitted 2021-05-23; First posted 2021-06-01 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Insomnia Chronic
Keywords: insomnia; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PEAR-003b PDT Intervention (Experimental): Participants will receive the PEAR-003b digital therapeutic, a Fitbit, and materials on sleep hygiene and healthy sleep tips. Using the Hugo platform, patient-generated engagement data, healthcare utilization, and patient activity/clinical outcomes for patients with insomnia will also be collected.
  Interventions: Device: PEAR-003b PDT Intervention; Device: Fitbit; Behavioral: Sleep education materials
- Control Arm (Placebo Comparator): Participants will receive a Fitbit, and materials on sleep hygiene and healthy sleep tips. Using the Hugo platform, patient-generated engagement data, healthcare utilization, and patient activity/clinical outcomes for patients with insomnia will also be collected.
  Interventions: Device: Fitbit; Behavioral: Sleep education materials

INTERVENTIONS:
Device: PEAR-003b PDT Intervention — The PEAR-003b digital therapeutic delivers CBT-I via mobile devices as 6 treatment core modules over 9 weeks.
  Arms: PEAR-003b PDT Intervention
Device: Fitbit — Patients will receive a Fitbit and receive standard of care
Behavioral: Sleep education materials — Patients will receive sleep hygiene and healthy sleep tips.

SUMMARY:
This will be a prospective multi-center controlled trial of 100 patients conducted to assess the real-world effectiveness of a mobile-delivered, prescription digital therapeutic (PDT) device delivering Cognitive Behavioral Therapy for Insomnia using a novel patient-centered data-sharing platform with linkage to Fitbit for 61 weeks

DETAILED DESCRIPTION:
This is a multi-center, randomized, controlled trial to assess the real-world effectiveness of a mobile-delivered, prescription digital therapeutic (PDT) device delivering Cognitive Behavioral Therapy for Insomnia (i.e., Somryst, herein called PEAR-003b) using a novel patient-centered data sharing platform (called Hugo), with linkage to Fitbit (Inspire 2), among 100 patients with chronic insomnia. Half of the patients with insomnia will receive the PEAR-003b digital therapeutic with linkage to the Hugo platform and Fitbit (Inspire 2) and half of the patients with insomnia will not receive the PDT but will receive a Fitbit and be enrolled in the Hugo platform. The treatment duration will be 9 weeks with a 21-, 35-, and 61-week follow-up. All patients will be evaluated at baseline, as well as prompted to complete additional assessments at weeks 9, 21, 35, and 61. The PEAR-003b intervention will deliver CBT-I via mobile devices as 6 treatment core modules over 9 weeks. Additionally, the Hugo platform will be used to collect patient-generated engagement data, healthcare utilization outcomes, and patient activity/clinical outcomes. These real-world data points and trends collected as part of this pilot investigation will help inform a future larger healthcare effectiveness and outcomes research study.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 22-64 years

  * English-speaking (both reading and writing in English required)
  * Diagnosis of chronic insomnia
  * Participant is willing and able to give consent and participate in study
  * Participant has an email account or is willing to create one and a smartphone able to download the necessary applications
  * Participant is willing and able to use the PDT, the Hugo data sharing platform and the syncable devices (e.g. Fitbit)
  * Participant has primary care at YNHH or Mayo Clinic

Exclusion Criteria:

* Pregnancy
* Shift work or family/other commitments that interfere with establishment of regular night-time sleep patterns, and if wake/sleep time is outside the ranges of 4:00h - 10:00h (wake time) and 20:00h - 02:00h (bed time)
* Absence of a reliable internet access and smartphone
* A reported diagnosis of psychosis, schizophrenia or bipolar disorder, or any medical disorders contraindicated with sleep restriction
* Current involvement in a non-medication treatment program for insomnia (participants are still eligible if they are taking traditional sleep medications)
* Those with untreated co-existing sleep conditions (e.g. sleep apnea)
* Those who have failed CBT for insomnia in the past

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S Ross, MD MHS, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Once the study has been completed, IPD will be shared in a way which will protect patient confidentiality using a data sharing platform for research purposes. The exact plan has yet to be decided.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available once the study has been completed

REFERENCES:
- [Derived] Dreyer RP, Berkowitz A, Yaggi HK, Schneeberg L, Shah ND, Emanuel L, Kolla B, Jeffery MM, Deeg M, Ervin K, Thorndike F, Ross JS. PreScription DigitaL ThErapEutic for Patients with Insomnia (SLEEP-I): a protocol for a pragmatic randomised controlled trial. BMJ Open. 2022 Aug 8;12(8):e062041. doi: 10.1136/bmjopen-2022-062041. PMID 35940841

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Started | 50 | 50
Completed | 47 | 49
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Participant Flow number differs from the Overall Number of Baseline Participants because two enrolled participants did not complete their baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | PEAR-003b PDT Intervention | Control Arm | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 enrolled participant did not answer this survey question
  years
    number analyzed (Participants) | 47 | 50 | 97
    (all) | 46.3 (12.09) | 43.9 (12.69) | 45.1 (12.40)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 35 | 34 | 69
  Male | 13 | 14 | 27
  Non-binary/third gender | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 43 | 43 | 86
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity
Description: Insomnia will be measured by the Insomnia Severity Index (ISI) score. Participants rate the severity of sleep problems (e.g. problems with sleep onset, sleep maintenance, and early morning awakening), interference with daytime functioning, how noticeable the impairment is to others, distress or concern caused by the sleep problem(s), as well as satisfaction with the current sleep pattern on a 5-point Likert scale. The ISI's total score ranges from 0 (not clinically significant) to 28 (clinically significant)
Time Frame: From baseline to 9 weeks post randomization
Population: Primary outcome measure was erased from study surveys and therefore not collected.
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Insomnia Severity
Description: as for outcome 1
Time Frame: From baseline to 21 weeks post-randomization
Population: The primary outcome measure was not asked in the study surveys and therefore not collected. As a result, this secondary outcome measure, a component of the primary outcome, cannot be calculated.
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Insomnia Severity
Description: as for outcome 1
Time Frame: From baseline to 35 weeks post-randomization
Population: as for outcome 2
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Insomnia Severity
Description: as for outcome 1
Time Frame: From baseline to 61 weeks post-randomization
Population: as for outcome 2
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Depressive Symptoms
Description: Depressive symptoms will be measured by the Patient Health Questionnaire (PHQ-8. The PHQ-8 is an 8 item 0 to 3 scale questionnaire. Total score ranges from 0 (not clinically significant) to 24 (clinically significant)
Time Frame: From baseline to 9 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 30
score on a scale | -2.0 [-4.0 to 0.0] | -1.5 [-5.0 to 1.0]

6. Secondary Outcome: Change in Depressive Symptoms
Description: as for outcome 5
Time Frame: From baseline to 21 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 20 | 30
score on a scale | -2.0 [-5.0 to 1.0] | -2.0 [-5.0 to 1.0]

7. Secondary Outcome: Change in Depressive Symptoms
Description: as for outcome 5
Time Frame: From baseline to 35 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 22 | 21
score on a scale | -2.0 [-4.0 to 1.0] | -4.0 [-8.0 to -1.0]

8. Secondary Outcome: Change in Depressive Symptoms
Description: as for outcome 5
Time Frame: From baseline to 61 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 23 | 21
score on a scale | -2.0 [-8.0 to 0.0] | 0.0 [-4.0 to 1.0]

9. Secondary Outcome: Change in Anxiety
Description: The General Anxiety Disorder-7 (GAD-7) is a widely used diagnostic self-report scale that screens, diagnoses, and assesses the severity of anxiety disorder. The GAD-7 is a 7-item 0 to 3 (0 = Not at all, 3 = Nearly every day) scale that measures the degree of severity of anxiety over the last 2 weeks with a total score ranging from 0 to 21, with a higher score indicating a more severe anxiety.
Time Frame: From baseline to 9 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 30
units on a scale | -2.0 [-5.0 to 1.0] | -1.0 [-2.0 to 1.0]

10. Secondary Outcome: Change in Anxiety
Description: as for outcome 9
Time Frame: From baseline to 21 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 20 | 30
score on a scale | -1.0 [-3.0 to 2.0] | -1.0 [-3.0 to 1.0]

11. Secondary Outcome: Change in Anxiety
Description: as for outcome 9
Time Frame: From baseline to 35 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 22 | 21
score on a scale | -1.0 [-3.0 to 2.0] | -1.0 [-4.0 to 0.0]

12. Secondary Outcome: Change in Anxiety
Description: as for outcome 9
Time Frame: From baseline to 61 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 23 | 21
score on a scale | -2.0 [-5.0 to 1.0] | -1.0 [-3.0 to 0.0]

13. Secondary Outcome: Change in Stress
Description: The Perceived Stress Scale (PSS) is a widely used self-reported 10-item questionnaire that assesses how stressful participants believe their life is. Scores range from 0 - 40 with higher scores pointing to more perceived stress.
Time Frame: From baseline to 9 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 30
score on a scale | -1.0 [-3.0 to 2.0] | -0.5 [-3.0 to 2.0]

14. Secondary Outcome: Change in Stress
Description: as for outcome 13
Time Frame: From baseline to 21 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 30 | 20
score on a scale | 0.0 [-2.0 to 3.0] | -1.5 [-4.0 to 1.0]

15. Secondary Outcome: Change in Stress
Description: as for outcome 13
Time Frame: From baseline to 35 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 22 | 21
score on a scale | -1.0 [-3.0 to 1.0] | -3.0 [-4.0 to 0.0]

16. Secondary Outcome: Change in Stress
Description: as for outcome 13
Time Frame: From baseline to 61 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 23 | 21
score on a scale | 0.0 [-3.0 to 3.0] | -1.0 [-4.0 to 1.0]

17. Secondary Outcome: Change in Quality of Life (PCS)
Description: Change in quality of life as measured in the Short Form 12 (SF-12). The physical health component (PCS) score ranges from 0-100 with higher scores representing better self-reported physical health.
Time Frame: From baseline to 9 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 30
score on a scale | -3.0 [-6.5 to 0.3] | -1.1 [-5.3 to 1.0]

18. Secondary Outcome: Change in Quality of Life (PCS)
Description: as for outcome 17
Time Frame: From baseline to 21 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 20 | 30
score on a scale | 0.5 [-4.3 to 4.8] | -2.6 [-7.2 to 1.4]

19. Secondary Outcome: Change in Quality of Life (PCS)
Description: as for outcome 17
Time Frame: From baseline to 35 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 22 | 21
score on a scale | -1.2 [-7.6 to 3.5] | -2.4 [-9.4 to 0.1]

20. Secondary Outcome: Change in Quality of Life (PCS)
Description: as for outcome 17
Time Frame: From baseline to 61 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 23 | 21
score on a scale | -1.0 [-5.0 to 3.8] | -4.1 [-8.3 to 0.4]

21. Secondary Outcome: Change in Daytime Sleepiness
Description: Daytime sleepiness is measured by the Epworth Sleepiness Scale (ESS) The ESS total score ranges from 0 (not clinically significant) to 24 (clinically significant)
Time Frame: From baseline to 9 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 30
score on a scale | -2.0 [-4.0 to 0.0] | 0.0 [-3.0 to 1.0]

22. Secondary Outcome: Change in Daytime Sleepiness
Description: as for outcome 21
Time Frame: From baseline to 21 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 20 | 30
score on a scale | -2.0 [-3.0 to -0.5] | 0.0 [-2.0 to 1.0]

23. Secondary Outcome: Change in Daytime Sleepiness
Description: as for outcome 21
Time Frame: From baseline to 35 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 22 | 21
score on a scale | 0.0 [-3.0 to 1.0] | -2.0 [-4.0 to 1.0]

24. Secondary Outcome: Change in Daytime Sleepiness
Description: as for outcome 21
Time Frame: From baseline to 61 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 23 | 21
score on a scale | -1.0 [-3.0 to 0.0] | 0.0 [-2.0 to 1.0]

25. Secondary Outcome: Healthcare Utilization
Description: Healthcare utilization will be reported as the number of outpatient visits with a primary care clinician or specialty care clinician.
Time Frame: From baseline to 9 weeks post-randomization
Population: The healthcare utilization outcomes data were not collected due to broken connections between the data aggregating platform and both the participant's wearable device and electronic health record. The team did not discover this until after the participant follow-up period concluded.
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Healthcare Utilization
Description: as for outcome 25
Time Frame: From baseline to 21 weeks post-randomization
Population: as for outcome 25
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Healthcare Utilization
Description: as for outcome 25
Time Frame: From baseline to 35 weeks post-randomization
Population: as for outcome 25
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Healthcare Utilization
Description: as for outcome 25
Time Frame: From baseline to 61 weeks post-randomization
Population: as for outcome 25
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Medication Utilization
Description: Medication utilization will be reported as the number of medication refills for sleep and/or psychotropic medications.
Time Frame: From baseline to 9 weeks post-randomization
Population: as for outcome 25
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Medication Utilization
Description: Medication utilization will be reported as the number of medication refills for sleep and/or psychotropic medications.
Time Frame: From baseline to 21 weeks post-randomization
Population: as for outcome 25
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Medication Utilization
Description: Medication utilization will be reported as the number of medication refills for sleep and/or psychotropic medications.
Time Frame: From baseline to 35 weeks post-randomization
Population: as for outcome 25
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Medication Utilization
Description: Medication utilization will be reported as the number of medication refills for sleep and/or psychotropic medications.
Time Frame: From baseline to 61 weeks post-randomization
Population: as for outcome 25
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Change in Sleep Efficiency
Description: Change in sleep efficiency, calculated as time spent sleeping divided by time spent in bed. This data is acquired from sleep diaries filled out by patient. (range 0-100 percentage points)
Time Frame: From baseline to 9 weeks post-randomization
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 38 | 35
percentage points | 14 (21.1) | 12.1 (11.5)

34. Secondary Outcome: Change in Sleep Efficiency
Description: as for outcome 33
Time Frame: From baseline to 21 weeks post-randomization
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 30
percentage points | 17.5 (12.7) | 13.8 (14.9)

35. Secondary Outcome: Change in Sleep Efficiency
Description: as for outcome 33
Time Frame: From baseline to 35 weeks post-randomization
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 24
percentage points | 14.9 (16.4) | 13.5 (15.8)

36. Secondary Outcome: Change in Sleep Efficiency
Description: as for outcome 33
Time Frame: From baseline to 61 weeks post-randomization
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 15 | 8
percentage points | 11.6 (15.6) | 15.8 (11.4)

37. Secondary Outcome: Change in Sleep Onset Latency
Description: Change in sleep-onset latency (SOL; hour), is based on the participants sleep diary and how many hours it took the participants to fall asleep.
Time Frame: From baseline to 9 weeks post-randomization
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 38 | 36
hours | 0.15 (2.21) | -0.193 (2.14)

38. Secondary Outcome: Change in Sleep Onset Latency
Description: as for outcome 37
Time Frame: From baseline to 21 weeks post-randomization
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 28 | 31
hours | -0.513 (2.058) | -0.765 (1.728)

39. Secondary Outcome: Change in Sleep Onset Latency
Description: as for outcome 37
Time Frame: From baseline to 35 weeks post-randomization
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 28 | 25
hours | -0.926 (1.729) | -0.94 (1.636)

40. Secondary Outcome: Change in Sleep Onset Latency
Description: as for outcome 37
Time Frame: From baseline to 61 weeks post-randomization
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 15 | 9
hours | -0.955 (1.35) | 0.184 (1.826)

41. Secondary Outcome: Change in Health Utility Score
Description: The Short Form 6 dimensions (SF-6D) is a health-related quality-of-life classification system that was developed from the SF-36 health survey (SF-36) and SF-12 health survey (SF-12). In this study, a scoring method was applied that focuses on seven of the health domains covered by the SF-12: Physical Functioning, Role Limitation (combined Physical and Emotional), Social Functioning, Bodily Pain, Mental Health, and Vitality- to create a single index of health. The resulting SF-6D is scored from 0.0 (worst measured health state) to 1.0 (best measured health state), with the difference being calculated to determine the change in health utility score for each arm in each time period. Data presented here is the percent change in score from baseline to 9 weeks post-randomization.
Time Frame: From baseline to 9 weeks post-randomization
Measure: Mean (Standard Error); unit: percent change
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 31
percent change | 1.7 (1.8) | -0.3 (1.3)

42. Secondary Outcome: Change in Health Utility Score
Description: The Short Form 6 dimensions (SF-6D) is a health-related quality-of-life classification system that was developed from the SF-36 health survey (SF-36) and SF-12 health survey (SF-12). In this study, a scoring method was applied that focuses on seven of the health domains covered by the SF-12: Physical Functioning, Role Limitation (combined Physical and Emotional), Social Functioning, Bodily Pain, Mental Health, and Vitality- to create a single index of health. The resulting SF-6D is scored from 0.0 (worst measured health state) to 1.0 (best measured health state), with the difference being calculated to determine the change in health utility score for each arm in each time period. Data presented here is the percent change in score from baseline to 21 weeks post-randomization.
Time Frame: From baseline to 21 weeks post-randomization
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 20 | 30
percentage change | 6.8 (3.1) | -1.6 (1.5)

43. Secondary Outcome: Change in Health Utility Score
Description: The Short Form 6 dimensions (SF-6D) is a health-related quality-of-life classification system that was developed from the SF-36 health survey (SF-36) and SF-12 health survey (SF-12). In this study, a scoring method was applied that focuses on seven of the health domains covered by the SF-12: Physical Functioning, Role Limitation (combined Physical and Emotional), Social Functioning, Bodily Pain, Mental Health, and Vitality- to create a single index of health. The resulting SF-6D is scored from 0.0 (worst measured health state) to 1.0 (best measured health state), with the difference being calculated to determine the change in health utility score for each arm in each time period. Data presented here is the percent change in score from baseline to 35 weeks post-randomization.
Time Frame: From baseline to 35 weeks post-randomization
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 22 | 21
percentage change | -3.8 (2.5) | 2.6 (1.8)

44. Secondary Outcome: Change in Health Utility Score
Description: The Short Form 6 dimensions (SF-6D) is a health-related quality-of-life classification system that was developed from the SF-36 health survey (SF-36) and SF-12 health survey (SF-12). In this study, a scoring method was applied that focuses on seven of the health domains covered by the SF-12: Physical Functioning, Role Limitation (combined Physical and Emotional), Social Functioning, Bodily Pain, Mental Health, and Vitality- to create a single index of health. The resulting SF-6D is scored from 0.0 (worst measured health state) to 1.0 (best measured health state), with the difference being calculated to determine the change in health utility score for each arm in each time period. Data presented here is the percent change in score from baseline to 61 weeks post-randomization.
Time Frame: From baseline to 61 weeks post-randomization
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 23 | 22
percentage change | 3.7 (2.8) | 0.5 (2.2)

45. Secondary Outcome: Change in Quality of Life (MCS)
Description: Change in quality of life as measured in the Short Form 12 (SF-12). The mental health component (MCS) score ranges from 0-100 with higher scores representing better self-reported mental health.
Time Frame: From baseline to 9 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 27 | 30
score on a scale | 2.2 [-0.4 to 8.1] | 3.0 [-1.2 to 6.8]

46. Secondary Outcome: Change in Quality of Life (MCS)
Description: as for outcome 45
Time Frame: From baseline to 21 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 20 | 30
score on a scale | 1.7 [-5.2 to 12.3] | 2.0 [-1.6 to 7.7]

47. Secondary Outcome: Change in Quality of Life (MCS)
Description: as for outcome 45
Time Frame: From baseline to 35 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 22 | 21
score on a scale | 3.2 [-5.4 to 6.4] | 5.7 [-1.0 to 9.9]

48. Secondary Outcome: Change in Quality of Life (MCS)
Description: as for outcome 45
Time Frame: From baseline to 61 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PEAR-003b PDT Intervention | Control Arm
Number analyzed (Participants) | 23 | 21
score on a scale | 1.9 [-2.9 to 6.7] | 2.2 [-2.5 to 10.8]

ADVERSE EVENTS:
Time Frame: up to 61 weeks post-randomization
Arm/Group | PEAR-003b PDT Intervention | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT04909229/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT04909229/ICF_001.pdf